CLINICAL TRIAL: NCT03452423
Title: The Effect on Gait Pattern in Patients Receiving Arthroscopic Cartilage Regeneration Facilitating Procedure (ACRFP) for Treatment of Osteoarthritis
Brief Title: The Effectiveness of Arthroscopic Cartilage Regeneration Facilitating Procedure for Patients With Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-XD41-074
Record Dates: First submitted 2018-02-01; First posted 2018-03-02 (Actual); Last update posted 2018-03-02 (Actual); Status verified 2017-11

CONDITIONS: Osteoarthritis of Knees
Keywords: Osteoarthritis of knees; Arthroscopic cartilage regeneration facilitating procedure (ACRFP); Foot pressure; Gait

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACRFP (Experimental): Patient suffering from osteoarthritis of knee joints, and planning to receive ACRFP, are enrolled into this study. Gait pattern is obtained preoperatively, 3 months, and 6 months postoperatively.
  Interventions: Procedure: ACRFP

INTERVENTIONS:
Procedure: ACRFP — Arthroscopic cartilage regeneration facilitating procedure (ACRFP) is a set of surgical procedures that combines resection of medial plica, medial and lateral capsular release, synovectomy of focal synovitis, and chondroplasty of loosened cartilage flaps as a rationale for the deliberate arthroscopic management of osteoarthritic knee.

SUMMARY:
The aim of this study is to discuss the effect of gait pattern in patients receiving arthroscopic cartilage regeneration facilitating procedure (ACRFP) for treatment of osteoarthritis of knees.

DETAILED DESCRIPTION:
Pain during gait is the most common and problematic symptom in individuals with osteoarthritis (OA) of knee joints. Limited range of motion, reduced walking speed, and a shortened stride length are also occasionally observed. These changes may be secondary or compensatory phenomena adopted by individuals to lessen the load on the OA-affected knees.

It is generally agreed that medial plica can produce symptoms in the knee joint, and can be successfully treated by arthroscopic resection when it becomes inflamed, thickened, and fibrotic. In 2006, Lyu and Hsu reported that medial plica had strong correlation with medial compartment osteoarthritis of knees. In their further studies disclosing the kinematic relationship of the medial plica with the medial femoral condyle found that medial plica might cause some degree of abrasion on the surface of medial femoral condyle during knee motion. The repeated injuries elicited by this abrasion phenomenon might trigger some inflammatory process to gradually damage the cartilage of knee.

Based on these findings, Lyu developed a concept of arthroscopic cartilage regeneration facilitating procedure (ACRFP) by arthroscopic resection of the medial plica, in addition to both medial and lateral capsular release, for the treatment of osteoarthritis of the knee joint. The clinical outcome of this procedure by eradication of the abrasion phenomenon caused by the tight, fibrotic, and hypertrophied medial plica, with decompression of the patellofemoral joint, the pain in most patients could be reduced, and the degenerative process in the medial compartment of some patients might be decelerated or arrested.

During the ACRFP, additional procedures such as synovectomy, abrasiochondroplasty, or partial menisectomy may also be carried out when necessary. It has been found that the elimination of the existing detrimental factors may provide a preferable environment for regeneration of the damaged cartilage.

Although the results of ACRFP for treatment of osteoarthritis of knee has been supported by several researches as being an effective method, it still lacks investigations on the gait pattern after such procedure. Therefore, the aim of this study is to discuss the effectiveness of the ACRFP for the patients with osteoarthritis of knee joints, specifically focused on their gait pattern.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages 20 and 85 who will receive ACRFP for treatment of osteoarthritis in the knee joints

Exclusion Criteria:

* Patients with walking disability

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-05-30 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Partial foot pressure as a percentage of body weight | Before intervention, at 3 months and 6 months after intervention
  ach footprint during gait are divided into 6 areas, which are medial forefoot, medial midfoot, medial hindfoot, lateral forefoot, lateral midfoot, and lateral hindfoot. The average partial foot pressure in each area was then calculated in terms of the percentage of body weight.

SECONDARY OUTCOMES:
The Knee injury and Osteoarthritis Outcome Score (KOOS) | Before surgery, at 3 months, and 6 months after intervention
  A questionnaire to assess the patient's subjective symptoms about their knee joints and associated problems caused by the disorders
Partial foot area as a percentage of body mass index (BMI) | Before surgery, at 3 months, and 6 months after intervention
  Each footprint during gait are divided into 6 areas, which are medial forefoot, medial midfoot, medial hindfoot, lateral forefoot, lateral midfoot, and lateral hindfoot. The average partial foot pressure in each area was then calculated in terms of the body mass index (BMI).
Gait Cadence | Before surgery, at 3 months, and 6 months after intervention
  The number of steps per minute
Walking speed | Before surgery, at 3 months, and 6 months after intervention
  The velocity of each single step
Single leg stance time | Before surgery, at 3 months, and 6 months after intervention
  The length of time of each foot at the stance phase
Step length | Before surgery, at 3 months, and 6 months after intervention
  The distance between the first point of contact of the foot with the ground and that of the contralateral foot
Step width | Before surgery, at 3 months, and 6 months after intervention
  The distance between the center of the heel contact and the following one, calculated perpendicularly to the direction of the horizontal axis drawn between the feet
Axis angle | Before surgery, at 3 months, and 6 months after intervention
  the angle formed by the medial tangent of the foot and the line from the second/third toe to the center of the heel

CONTACTS AND LOCATIONS:
Overall Officials: Shuo-Suei Hung, PhD, Principal Investigator — Buddhist Taipei Tzu Chi General Hospital
Locations (1):
- Buddhist Taipei Tzu Chi General Hospital, New Taipei City, Taiwan